CLINICAL TRIAL: NCT06212778
Title: Relationship Between Nutritional Status, Hand Grip Strength, and Fatigue in Hospitalized Older Adults With Type 2 Diabetes Mellitus.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202309041RINB
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As the proportion of the elderly population increases, so does the number of people suffering from diabetes mellitus (DM). Fatigue is common in elderly patients with type 2 diabetes, and malnutrition may lead to a decrease in muscle strength, thereby aggravating their fatigue symptoms; however, there is still a lack of relevant research on this group in Taiwan. Therefore, the purposes of this study are to understand the current status and correlation of basic attributes, nutritional status, handgrip strength and fatigue in hospitalized older adults with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus (DM)is increasing among the elderly population in Taiwan, and fatigue is a common troublesome symptom that likely impacts their quality of life and diabetes self-management. Malnutrition is one of the causes of fatigue symptoms in the elderly, and the worse the nutritional status, the worse the hand grip strength performance; the better the grip strength performance, the lower the degree of fatigue symptoms. It can be inferred that the worse the nutritional status, the worse the handgrip strength, which will in turn have an aggravating impact on fatigue symptoms. According to previous literature, handgrip strength may be an important mediating variable between nutritional status and fatigue. However, there are still no relevant studies on hospitalized older adults with type 2 diabetes mellitus.

Therefore, the purposes of this study are to: (1) understand the basic attributes, nutritional status, handgrip strength and fatigue symptoms in hospitalized older adults with type 2 diabetes mellitus. (2) explore the correlation between nutritional status, handgrip strength and fatigue symptoms in hospitalized older adults with type 2 diabetes mellitus, so as to serve as a reference for future clinical care to improve fatigue in elderly patients with type 2 diabetes mellitus.

This study adopted a cross-sectional, correlational design, using structured questionnaires and a Camry Digital Handgrip Dynamometer to collect data. Participants will be recruited from a metabolism & endocrinology ward at a medical center in northern Taiwan using purposive sampling. The Chinese version of a structured questionnaire, including the demographic and clinical characteristic form, the Mini Nutritional Assessment , and the Fatigue Symptom Inventory will be used. A sample of 54 participants with type 2 diabetes mellitus will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* People who are aged 60 or above
* Diagnosed with type 2 diabetes mellitus
* Conscious and agree to participate in the study.

Exclusion Criteria:

* People who have a cognitive impairment or unable to communicate
* Unable to use the handgrip dynamometer with their dominant hand
* Under active treatment for cancer.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized older adults with type 2 diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 30 mins
  Fatigue Symptom Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan